CLINICAL TRIAL: NCT04011644
Title: Integrating mHealth for Alcohol Use Disorders Into Clinical Practice
Brief Title: Mobile Health for Alcohol Use Disorders in Clinical Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0337; R01AA024150 (NIH); A532007 (Other: UW Madison); SMPH/FAMILY MED/RES GRANTS (Other: UW Madison); Protocol Version 8/18/2021 (Other: UW Madison)
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Results first posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Alcohol Drinking; Telemedicine
Keywords: implementation; alcohol drinking; mHealth; wellness
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: The study will have rolling enrollment over two years. Patients will be enrolled and randomized to one of three interventions for 12 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Self monitored (Active Comparator): Patients of this group will continue receiving regular care from their physician with no interference from the two experimental groups. Patient subjects will download the app on their Android or Apple smart phone that will direct them to external information hosted on the internet that may help reduce their drinking (e.g., NIAAA resources). For the first 12 weeks, once a week patients can set a weekly goal related to their alcohol use or other health related behaviors (e.g., "I will only drink on Friday this week."). At the end of the week subjects will be prompted to take a weekly survey, which will include questions such as a variation of the brief alcohol monitor (BAM) and timeline followback. Patients will then receive feedback on the amount of drinks they had compared to their goal. Then the patient will set a new goal for the following week. Patients will complete quarterly surveys on the A-CHESS app to assess study outcomes.
  Interventions: Behavioral: A-CHESS self-monitored
- Peer supported (Experimental): Patients will be asked to take the same surveys and have the access to the same information as the self-monitoring group. Patient subjects in this group will have access to discussion boards where they can talk to one another and have the ability to share and see stories of other patients. The only involvement of someone other than patients themselves in the peer-supported group will be by a sponsor (i.e., a dedicated user from the area with a sustained history of successful alcohol reduction). The sponsor will participate in discussion groups and encourage use of the system. Patient-reported feedback will be presented directly to the patient.
  Interventions: Behavioral: A-CHESS peer-supported
- Clinically integrated (Experimental): Patients in the clinically integrated group will receive the same intervention as the peer-supported group aside from three differences: 1) patients have the option to share selected elements of their app data with the University of Wisconsin (UW) Health health coach, 2) the health coach will replace the role of the sponsor in the peer-support group, and 3) patients will have the option to attend an initial 60- to 90-minute and two 30-minute follow-up consultations with the health coach in-person, via phone, or via video chat.
  Interventions: Behavioral: A-CHESS clinically-integrated

INTERVENTIONS:
Behavioral: A-CHESS self-monitored — Patients have access to a smart phone app that provides information on tips on how to reduce drinking, a drink tracker, a journal, discussion boards, and private messaging with a research team member. Patients set weekly goals related to their drinking, reassess each week, and set a new goal for the upcoming week.
  Arms: Self monitored
Behavioral: A-CHESS peer-supported — Patients have access to a smart phone app that provides information on tips on how to reduce drinking, a drink tracker, a journal, discussion boards, and private messaging with a counselor. Patients set weekly goals related to their drinking, reassess each week, and set a new goal for the upcoming week.
  Arms: Peer supported
Behavioral: A-CHESS clinically-integrated — Patients have access to a smart phone app that provides information on tips on how to reduce drinking, a drink tracker, a journal, discussion boards, and private messaging with a health coach. Patients set weekly goals related to their drinking, reassess each week, and set a new goal for the upcoming week.
  Arms: Clinically integrated

SUMMARY:
This study evaluates the impact on risky drinking days and quality of life for patients with alcohol use disorder among patients who use a mobile health smart phone application. A third of the participants will receive access to the smart phone app without any monitoring; a third of the participants will receive access to the smart phone app monitored by and connected with a peer mentor; a third will receive access to the smart phone app monitored by and connected with a health coach who works within a healthcare system.

DETAILED DESCRIPTION:
Patients in the trial will be given versions of an evidence-based mobile-health (mHealth) system (re-design based on A-CHESS) that is delivered using different implementation strategies according to study group. A-CHESS has more than 18 services designed to improve social relatedness, coping competence, and intrinsic motivation. The following describes key A-CHESS services that will be tested in the current study:

* Welcome message - patients write why they are choosing to reduce their drinking.
* Coping with Cravings - the system automatically notifies nearby pre-approved friends, family, and peers, who can respond to a request for support. The patient can also be linked to positive activities, such as suggested games to download and play and audio/video-based relaxation recordings.
* Monitoring functionality- self-assessment measures, record of A-CHESS use, and prediction of the patient's likelihood of having a heavy drinking episode in the next week. A-CHESS sends patients with worrisome responses suggestions of coping skills, online peer support, healthy events, etc. With patient permission, a prediction of high-risk can be shared with others in a position to provide support.
* Triage and feedback functionality is designed to derail a setback in goal attainment, giving the patient 'just in time,' tailored support by linking patients to relevant A-CHESS resources or individuals (depending on group assignment).
* The Specialist Report, harvests clinically relevant data from A-CHESS and presents it to a peer mentor (in the peer-supported group) or a health coach (in the clinically integrated group), at which point they may intervene with patients (e.g., through texting in A-CHESS).
* Facilitated discussion groups (in the clinically integrated group.) Discussions are monitored daily by an A-CHESS coach.
* Library - information about healthy lifestyle choices, calendar of healthy events in the area, etc.
* Drink tracker and report feature - patients to self-monitor their drinking and each week see a summary of how they did the past week.
* Profiles about why patients want to reduce their drinking.

All patients enrolled in the study will participate in a 3-month intervention period followed by a 9-month follow-up period, for a total of 12 months. All patient will undergo a 72-hour run-in period. After 72 hours, patients who remain in the study will be randomized to one of the following groups and receive the appropriate access to features. One group will operate independently; one group will have help from a peer-mentor; one group will be connected to a healthcare system by a health coach.

ELIGIBILITY:
Inclusion Criteria:

* are 21+ years old,
* interested in learning about ways to reduce drinking,
* willing to download and use A-CHESS,
* lives in within the geographical boundaries of the UW Health system
* be able to understand and sign an electronic consent form in English,
* own an Apple or android smart phone,
* meets the criteria for at risk drinking on the AUDIT screening,
* responds yes to at least one question on the Alcohol Use Disorder (AUD) Diagnostic and Statistical Manual-5 survey, and
* indicates in the past week they have had at least 7 drinks and 3 on a single day (women), or had at least 14 drinks and 4 on a single day (men).

Exclusion Criteria:

* has a severe alcohol use disorder (yes to 6+ items on the Alcohol Use Disorder (AUD) Diagnostic and Statistical Manual-5)
* have a current psychotic disorder
* have an acute medical problem requiring immediate hospitalization
* have a known terminal illness

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2020-03-23 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Quanbeck, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UW Health at the American Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data collected during the trial, after deidentification will be available to researchers for independent verification of study outcomes or to conduct subsequent clinical research, whose proposed use of the data has been approved by an independent review committee identified for this purpose.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Beginning 9 months after publication of primary outcomes, and ending 3 years following publication.
Access Criteria: Proposals should be directed to PI Andrew Quanbeck at arquanbe@wisc.edu. If approved after review by regulatory counsel, requestors will enter into a formal data sharing agreement. Data will be shared via encrypted single-user file transmission protocol.

REFERENCES:
- [Derived] Quanbeck A, Chih MY, Park L, Li X, Xie Q, Pulvermacher A, Voelker S, Lundwall R, Eby K, Barrett B, Brown R. A randomized trial testing digital medicine support models for mild-to-moderate alcohol use disorder. NPJ Digit Med. 2024 Sep 14;7(1):248. doi: 10.1038/s41746-024-01241-2. PMID 39271938
- [Derived] Park LS, Chih MY, Stephenson C, Schumacher N, Brown R, Gustafson D, Barrett B, Quanbeck A. Testing an mHealth System for Individuals With Mild to Moderate Alcohol Use Disorders: Protocol for a Type 1 Hybrid Effectiveness-Implementation Trial. JMIR Res Protoc. 2022 Feb 18;11(2):e31109. doi: 10.2196/31109. PMID 35179502

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A three-pronged recruitment strategy encompassing clinical settings, community-based organizations, and public media was used. Clinical study champions, including primary care providers, behavioral health specialists, etc., provided information to potentially eligible patients. Leaders from underrepresented communities promoted the study to their respective diverse populations. Lastly, targeted digital, television, and print media promoted the study broadly.
Pre-assignment Details: The site staff were not enrolled in the clinical trial that is represented in the overall study flow diagram above and as such are not included in it. They were engaged in a post hoc interview to understand the study results for an exploratory analysis.
Period: Overall Study
Arm/Group | Self Monitored | Peer Supported | Clinically Integrated
Started | 185 | 186 | 187
Completed | 139 | 132 | 102
Not Completed | 46 | 54 | 85

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Self Monitored | Peer Supported | Clinically Integrated | Total
Number analyzed (Participants) | 185 | 186 | 187 | 558
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.80 (12.9) | 42.8 (12.9) | 42.6 (12.9) | 42.8 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 122 | 123 | 365
  Male | 65 | 64 | 64 | 193
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 4 | 14
  Not Hispanic or Latino | 181 | 180 | 183 | 544
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 0 | 3
  Asian | 5 | 2 | 4 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 2
  Black or African American | 7 | 8 | 10 | 25
  White | 170 | 167 | 170 | 507
  More than one race | 0 | 3 | 1 | 4
  Unknown or Not Reported | 1 | 4 | 1 | 6
Education [Count of Participants; unit: Participants]
  < High school | 0 | 2 | 1 | 3
  HS or GED | 16 | 19 | 32 | 67
  Vocation or associate | 35 | 34 | 16 | 85
  Bachelors | 76 | 83 | 76 | 235
  Masters | 44 | 29 | 48 | 121
  Doctorate | 14 | 19 | 14 | 47
AUDIT Category [Count of Participants; unit: Participants]
  Low risk | 39 | 53 | 41 | 133
  Harmful drinking | 85 | 72 | 84 | 241
  Alcohol dependence | 61 | 61 | 62 | 184
Percentage of heavy drinking days (PHDD) [Mean (Standard Deviation); unit: percentage] — One participant in the Clinically Integrated group did not submit baseline measures for PHDD, QOL-PH, and QOL-MH, so the sample size for this group and these outcomes was 186, not the original number, 187.
  In the baseline and follow-up surveys, the participants were asked to report the number of risky drinking days in the last 7 days. The Percentage of Heavy Drinking Days (PHDD) was calculated by dividing the number of reported risking drinking days by 7. Population: One participant in the Clinically Integrated group did not submit baseline measures for PHDD, QOL-PH, and QOL-MH, so the sample size for this group and these outcomes was 186, not the original number, 187.
  percentage
    number analyzed (Participants) | 185 | 186 | 186 | 557
    (all) | 37.1 (30.6) | 36.2 (31.2) | 41.9 (31.4) | 38.4 (31.1)
Quality of life-physical health, QOL-PH [Mean (Standard Deviation); unit: T-score] — The Quality-of-Life Physical Health (QoL-PH) was measured using the four global physical health survey items in the Patient-Reported Outcome Measurement Information System (PROMIS) global health short form (SF10 ver.1.2). The raw scores for physical health (range: 4 to 20) were converted to T-scores (range: 16.2 to 67.7) using the PROMIS scoring manual (p.16). T-scores reported here are standardized scores that can be compared to the US general population and have a mean QOL score of 50 with a standard deviation of 10. Higher scores mean better physical health. Population: One participant in the Clinically Integrated group did not submit baseline measures for PHDD, QOL-PH, and QOL-MH, so the sample size for this group and these outcomes was 186, not the original number, 187.
  T-score
    number analyzed (Participants) | 185 | 186 | 186 | 557
    (all) | 48.4 (6.3) | 48.1 (6.7) | 48.3 (6.5) | 48.3 (6.5)
Quality of life-mental health, QOL-MH [Mean (Standard Deviation); unit: T-scores] — The Quality-of-Life Mental Health (QoL-MH) was measured using the four global mental health survey items in the Patient-Reported Outcome Measurement Information System (PROMIS) global health short form (SF10 ver.1.2). The raw scores for mental health (range: 4 to 20) were converted to T-scores (range: 21.2 to 67.6) using the PROMIS scoring manual (p.16). T-scores reported here are standardized scores that can be compared to the US general population and have a mean QOL score of 50 with a standard deviation of 10. Higher scores mean better mental health. Population: One participant in the Clinically Integrated group did not submit baseline measures for PHDD, QOL-PH, and QOL-MH, so the sample size for this group and these outcomes was 186, not the original number, 187.
  T-scores
    number analyzed (Participants) | 185 | 186 | 186 | 557
    (all) | 45.5 (6.9) | 45.5 (7.5) | 45.4 (6.9) | 45.4 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Heavy Drinking Days, PHDD
Description: Percentage of self-reported Heavy Drinking Days (HDD: 5 or more standard drinks on any day for men under 65, 4 or more standard drinks for women and men over 65) in the last 7 days
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: percentage of heavy drinking days
Arm/Group | Self Monitored | Peer Supported | Clinically Integrated
Number analyzed (Participants) | 139 | 130 | 100
percentage of heavy drinking days | 24.4 (28.2) | 21.4 (28.9) | 21.3 (30.4)
Statistical Analysis 1: Comparison: Self Monitored vs Peer Supported vs Clinically Integrated; Test type: Superiority; p = 0.688, Mixed Models Analysis; Quanbeck,A.et al. A randomized trial testing digital medicine support models for mild-to-moderate alcohol use disorder. npj Digit. Med.7,248(2024)

2. Primary Outcome: Quality of Life-Physical Health
Description: The physical health subscale of Patient Reported Outcomes Measurement Information System (PROMIS) Global-10 short form was used to assess the quality of life-physical health (QoL-PH). It consists of 4 questions that assess overall physical health aspect of quality of life. Each question will ask patients to indicate their physical health on a scale of 1 (poor) to 5 (excellent). The raw scores of physical health scores (range: 0 to 20) are converted to T-scores (16.2 to 67.7). Higher scores mean better physical health aspects of quality of life.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: T-Scores
Arm/Group | Self Monitored | Peer Supported | Clinically Integrated
Number analyzed (Participants) | 139 | 130 | 100
T-Scores | 48.5806 (6.81051) | 49.2869 (6.44004) | 48.1010 (7.45609)
Statistical Analysis 1: Comparison: Self Monitored vs Peer Supported vs Clinically Integrated; Test type: Superiority; p = 0.261, Mixed Models Analysis

3. Primary Outcome: Quality of Life-Mental Health
Description: The mental health subscale of Patient Reported Outcomes Measurement Information System (PROMIS) Global-10 short form was used to assess the quality of life-mental health (QoL-MH). It consists of 4 questions that assess overall mental health aspect of quality of life. Each question will ask patients to indicate their mental health on a scale of 1 (poor) to 5 (excellent). The raw scores of mental health scores (range: 0 to 20) are converted to T-scores (21.2 to 67.6). Higher scores mean better mental health aspects of quality of life.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: T-Scores
Arm/Group | Self Monitored | Peer Supported | Clinically Integrated
Number analyzed (Participants) | 139 | 130 | 100
T-Scores | 46.7439 (8.25969) | 47.6715 (8.30113) | 48.1160 (7.03693)
Statistical Analysis 1: Comparison: Self Monitored vs Peer Supported vs Clinically Integrated; Test type: Superiority; p = 0.014, Mixed Models Analysis

4. Secondary Outcome: Number of Patients Who Are Willing to Share Data
Description: Patients in the clinically-integrated arm will have the option to share their data collected by A-CHESS with the health coach. Knowing how many patients are willing to share data about their drinking will allow researchers to make hypotheses about how effective A-CHESS can be in a healthcare setting. We did not collect data for this metric.
Time Frame: 12 months
Population: We did not collect data for this metric.
Arm/Group | Self Monitored | Peer Supported | Clinically Integrated
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Number of Hospital Nights in the Past 6 Months
Description: Patients will be asked to indicate hospital stay (nights) in the past 6 months. Researchers will include this in the cost-effectiveness analysis.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Hospital nights
Arm/Group | Self Monitored | Peer Supported | Clinically Integrated
Number analyzed (Participants) | 131 | 128 | 101
Hospital nights | 0.0534 (0.35762) | 0.0469 (0.39404) | 0.2178 (1.34613)
Statistical Analysis 1: Comparison: Self Monitored vs Peer Supported vs Clinically Integrated; A univariate analysis (Analysis of Covariance or ANCOVA) was conducted to compare the number of hospital days among the three groups controlling for baseline assessment of the dependent variable and design factors (i.e., Sex and Severity); Test type: Superiority; p = 0.908, ANCOVA

6. Secondary Outcome: Cost of Implementation of Each Intervention Arm in US Dollars
Description: The cost (in US dollars) of the intervention will be calculated to determine cost-effectiveness of the study.
Time Frame: up to 3 years
Population: Cost reflects total number enrolled, not number completed, to account for program being at full capacity.
Measure: Number; unit: dollars
Arm/Group | Self Monitored | Peer Supported | Clinically Integrated
Number analyzed (Participants) | 185 | 186 | 187
dollars | 0 | 71750 | 124250

7. Secondary Outcome: Score of Alcohol Use Disorders Identification Test (AUDIT) Screening Tool
Description: The Alcohol Use Disorders Identification Test (AUDIT) screening tool was used to assess patient alcohol severity. The screening tool consists of 10 questions with 5 possible answers (scoring 0-4). The sum scores of the 10 items are the scale scores ranging from 0 to 40. Higher scores indicate greater alcohol severity.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Self Monitored | Peer Supported | Clinically Integrated
Number analyzed (Participants) | 132 | 127 | 99
Scores on a scale | 9.0303 (4.91289) | 9.3386 (5.9271) | 8.8283 (5.54948)
Statistical Analysis 1: Comparison: Self Monitored vs Peer Supported vs Clinically Integrated; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.206, ANCOVA

8. Secondary Outcome: Score of the Diagnostic and Statistical Manual- 5 Alcohol Use Disorder (AUD) Severity
Description: The Diagnostic and Statistical Manual of Mental Disorders 5th edition criteria of alcohol use disorder will be used to assess the patient's alcohol use disorder severity. Each item has a score of 1 for agreement or 0 for disagreement of a statement. The sum score of all 11 items is the scale score (range of 0-11 - higher scores indicate greater severity). The severity of the AUD can also be defined as 1) mild: 2 to 3 symptoms; 2) moderate: 4 to 5 symptoms; 3) severe: 6+ symptoms.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Self Monitored | Peer Supported | Clinically Integrated
Number analyzed (Participants) | 110 | 109 | 71
Scores on a scale | 2.5364 (1.76447) | 2.5229 (1.65326) | 2.9178 (2.17763)
Statistical Analysis 1: Comparison: Self Monitored vs Peer Supported vs Clinically Integrated; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.104, ANCOVA

9. Secondary Outcome: Score of Relatedness as Assessed by the CHESS Bonding Scale
Description: The study will assess how connected patients feel with others. Greater connectedness is associated with fewer risky drinking days. Patients are asked five Likert-scale questions about their relationships with others, responding on a 1-5 scale from 'Never' to 'Nearly Always.' Mean scores are calculated as scale scores, ranging from 1 to 5. Higher scores indicate greater perceived relatedness with others.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Scores
Arm/Group | Self Monitored | Peer Supported | Clinically Integrated
Number analyzed (Participants) | 139 | 130 | 100
Scores | 2.3022 (0.85985) | 2.7538 (0.87037) | 2.668 (0.95525)
Statistical Analysis 1: Comparison: Self Monitored vs Peer Supported vs Clinically Integrated; Test type: Superiority; p < 0.001, Mixed Models Analysis

10. Secondary Outcome: Score of Competence as Assessed by the Perceived Competence Scale (PCS)
Description: The study will assess patients' perceptions of their ability to control and reduce their drinking in order to meet their alcohol use goals. Patients tend to drink less when they feel more confident in managing their alcohol use. Patients will respond to four questions from the Perceived Competence Scale (PCS) about their confidence in responsibly managing alcohol use in various situations. Responses are on a 1-7 scale, from 'Not at all' to 'Very true.' Mean scores (ranging from 1 to 7) are used as the scale scores, with higher scores indicating greater confidence in controlling or reducing drinking.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Scores
Arm/Group | Self Monitored | Peer Supported | Clinically Integrated
Number analyzed (Participants) | 138 | 130 | 87
Scores | 5.1377 (1.26652) | 5.0788 (1.34071) | 5.39 (1.50013)
Statistical Analysis 1: Comparison: Self Monitored vs Peer Supported vs Clinically Integrated; Test type: Superiority; p = 0.025, Mixed Models Analysis

11. Secondary Outcome: Score of Autonomous Motivation as Assessed by Revised Treatment Self Regulation Questionnaire
Description: The study assesses how motivated patients are by their own goals. Patients typically drink less when they, themselves, want to reduce their alcohol. Patients will be asked 6 questions from the autonomous motivation subscale of the Treatment Self-Regulation Questionnaire (TSRQ) about why they will reduce their alcohol use and can indicate how much they identify with each statement on a 1-5 scale corresponding to "Not true" to "Very true", respectively. The mean scores are the scale scores, ranging from 1 to 5. Higher scores mean more autonomous motivation to control and reduce alcohol use.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Scores
Arm/Group | Self Monitored | Peer Supported | Clinically Integrated
Number analyzed (Participants) | 138 | 130 | 100
Scores | 3.8913 (0.67081) | 3.9244 (0.7311) | 4.0283 (0.811)
Statistical Analysis 1: Comparison: Self Monitored vs Peer Supported vs Clinically Integrated; Test type: Superiority; p = 0.555, Mixed Models Analysis

12. Secondary Outcome: Time of Tula Used
Description: The time that participants spent using Tula will be assessed.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Self Monitored | Peer Supported | Clinically Integrated
Number analyzed (Participants) | 185 | 186 | 187
Seconds | 17142.98 (15043.75) | 19851.64 (16160.12) | 17000.83 (12961.23)
Statistical Analysis 1: Comparison: Self Monitored vs Peer Supported vs Clinically Integrated; Test type: Superiority; p = 0.131, Kruskal-Wallis

13. Secondary Outcome: Number of Setback Status Triggered by A-CHESS
Description: The patient's ability to meet their weekly goal will be assessed. When patients are not on track to meet their weekly goal a setback alert will be triggered.
Time Frame: 12 months
Population: We did not implement this setback alert so no data are collected for this measure.
Arm/Group | Self Monitored | Peer Supported | Clinically Integrated
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Variables Used for Predictive Setback Status
Description: The variables that help predict a setback will be assessed and reported. Knowing the variables for setbacks will help researchers program A-CHESS to better predict when patients are likely to have a setback.
Time Frame: up to 3 years
Population: We did not implement this setback alert so no data are collected for this measure.
Arm/Group | Self Monitored | Peer Supported | Clinically Integrated
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Number of Response Statuses Addressed
Description: Clinicians and patients will be alerted when the system predicts that they may have a setback. This allows researchers to know how useful patients and health coaches found the alerts.
Time Frame: up to 3 years
Population: We did not implement this setback alert so no data are collected for this measure.
Arm/Group | Self Monitored | Peer Supported | Clinically Integrated
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Pages Viewed on A-CHESS
Description: The number of pages viewed by patients and health coaches will be assessed know how useful patients found different content.
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: Page view counts
Arm/Group | Self Monitored | Peer Supported | Clinically Integrated
Number analyzed (Participants) | 185 | 186 | 187
Page view counts | 753.12 (517.05) | 891.84 (544.44) | 773.1 (458.18)
Statistical Analysis 1: Comparison: Self Monitored vs Peer Supported vs Clinically Integrated; Test type: Superiority; p = 0.02, Kruskal-Wallis

17. Secondary Outcome: Number of Patient Protection Factors Assessed by a Revised Brief Alcohol Monitor
Description: Patients will take a revised Brief Alcohol Monitor survey weekly that asks patients to indicate whether any of the five protection factors exist (sleep, mood, social interaction, work, and urges to drink). The protective factor score is the sum of the number of protection factor items reported by patients during the study period. The scores of the protective factors were planned to be used in the lapse prediction model. Since the study plan changes and the lapse prediction was not the focus of the study, only descriptive statistics are reported. No additional statistical analysis was conducted. Scores range from 7-35. Lower scores indicate a worse outcome for each factor.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Self Monitored | Peer Supported | Clinically Integrated
Number analyzed (Participants) | 113 | 113 | 73
Score on a scale | 21.96 (5.45) | 23.02 (5.25) | 23.48 (5.63)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Self Monitored | Peer Supported | Clinically Integrated
All-Cause Mortality (participants affected / at risk) | 0/185 | 0/186 | 0/187
Serious Adverse Events (participants affected / at risk) | 0/185 | 0/186 | 0/187
Other Adverse Events (participants affected / at risk) | 0/185 | 0/186 | 0/187

LIMITATIONS AND CAVEATS:
Use of convenience sampling may limit generalizability to other populations; The study did not include a pure control group since doing so would require a "sham device," which was deemed impractical; The study took place during the COVID pandemic, where drinking rates increased nationwide including in Wisconsin.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-13): https://cdn.clinicaltrials.gov/large-docs/44/NCT04011644/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-09): https://cdn.clinicaltrials.gov/large-docs/44/NCT04011644/ICF_001.pdf